CLINICAL TRIAL: NCT04026451
Title: Use of Spectral Analysis of Electroencephalographic Activity to Guide Deep Sedoanalgesia and Its Effect on Propofol Consumption in Patients Hospitalized in the Intensive Care Unit: a Pilot Study
Brief Title: Spectral Edge Frequency From Spectral EEG Analysis to Guide Deep Sedation in the Critical Care Setting (Pilot)
Acronym: SEFICU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was suspendend because the protocol and the aims were modified
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Antonello Penna, Anesthesiologist, MD, PhD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1009/18
Record Dates: First submitted 2019-07-15; First posted 2019-07-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Deep Sedation; Mechanical Ventilation
Keywords: Sedation; EEG; Mechanical Ventilation; Critical Care; Propofol
MeSH Terms: interventions — Deep Sedation; Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Critical care patients with an indication of deep sedation and mechanical ventilation will be sedated with an infusion of propofol and fentanyl guided by SEF95 obtained by SedLine® monitor to keep a SAS 1-2. The target of SEF95 will be 10-13 Hz to keep SAS 1-2.
  Interventions: Device: Sedation guided by SEF95 (10-13 Hz) from SedLine® monitor; Behavioral: Sedation guided by SAS scale (1-2); Drug: Deep sedation with propofol andfentanyl; Procedure: Mechanical Ventilation
- Control (Active Comparator): Critical care patients with an indication of deep sedation and mechanical ventilation will be sedated with an infusion of propofol and fentanyl guided by SAS (1-2). SedLine® monitor will be also used in these patients but the screen will be covered.
  Interventions: Behavioral: Sedation guided by SAS scale (1-2); Drug: Deep sedation with propofol andfentanyl; Procedure: Mechanical Ventilation

INTERVENTIONS:
Device: Sedation guided by SEF95 (10-13 Hz) from SedLine® monitor — Dosage of propofol and fentanyl will be guided by SEF95 value between 10-13 Hz. If SEF95 is lower than 10 Hz, the infusion rate of propofol and fentanyl will be diminished; if SEF95 is higher than 13 Hz, the infusion rate of propofol and fentanyl will be increased; and if SEF95 is between 10-13 Hz, then the infusion rate will be kept.
  Arms: Intervention
Behavioral: Sedation guided by SAS scale (1-2) — Dosage of propofol and fentanyl will be guided by SAS to keep a value of 1-2. If SAS is higher than 1-2, then the infusion rate of propofol and fentanyl will be increased; and if SAS is 1-2, then the infusion rate of propofol and fentanyl will be maintained.
Drug: Deep sedation with propofol andfentanyl — Propofol and fentanyl will be infused to reach a score in the SAS of 1-2
Procedure: Mechanical Ventilation — Critically ill patients will be ventilated mechanically following the clinical indication.

SUMMARY:
Critically ill patients under mechanical ventilation (MV) have pain, anxiety, sleep deprivation and agitation. The use of analgesics and sedatives drugs (sedoanalgesia) is a common practice to produce pain relief and comfort during the VM. Despite its usefulness, it has been documented that the excessive use of sedatives is associated with an increased risk of prolonging the stay under MV and in the Intensive Care Unit (ICU). To avoid this, current evidence suggests the use of protocols guided to clinical goals, such as the sedation-agitation scale (SAS), or daily suspension of infusions to avoid excess sedation. These protocols minimize the prescription of deep sedation, which is still necessary for 20-30% of patients.

Monitoring of sedation with electroencephalography in the ICU has been underutilized. In fact, only the use of indices that are generated from algorithms of the electroencephalographic signal processing has been reported. However, it has been shown that the use of these monitoring systems does not benefit the heterogeneous groups of patients in MV. Currently, the clinical monitors used to measure the effect of drugs used in a sedoanalgesia show in the screen the spectrogram of the brain electrical signal and quantify the frequency under which 95% of the electroencephalographic power is located, known as spectral edge frequency 95 (SEF95). This value in a person who is conscious is usually greater than 20 Hz, in a patient undergoing general anesthesia it is between 10 and 15 Hz. In preliminary measurements, in deeply sedated patients in the ICU, SEF95 values are under 5 Hz. This would indicate that patients in the ICU are being overdosed. It is unknown if in cases with an indication of deep sedation, the use of monitoring by spectrogram is superior to the standard management guided at clinical scales, such as SAS.

Therefore, the investigators propose the following hypothesis: In patients with an appropriate indication of deep sedation (SAS 1-2), the sedoanalgesia guided by the spectral edge frequency 95 reduces the consumption of propofol compared to the deep sedoanalgesia guided by the sedation scale agitation in MV patients in the ICU maintaining a clinically adequate level of sedation.

DETAILED DESCRIPTION:
To determine whether deep sedoanalgesia guided by the spectral edge frequency 95 decreases propofol consumption with respect to deep sedoanalgesia guided by the sedation-agitation scale in patients hospitalized in the Intensive Care Unit under mechanical ventilation.

* Group intervention: sedation will be guided by SEF95 and SAS. Patients will be sedated to keep a SAS 1-2 with a SEF95 between 10 to 13 Hz.
* Group control: sedation will be guided by SAS. However, SEF95 will be also recorded but covered.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Indication of deep sedation with propofol and fentanyl for more than 48 h

Exclusion Criteria:

* Brain damage
* Cognitive impairment
* Allergy to propofol or fentanyl
* Limitation of therapeutic effort
* Liver chronic disease Child C
* Prone positioning and use of neuromuscular blocking agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of propofol | 48 hours
  It will be measured using HPLC

SECONDARY OUTCOMES:
Total dose of propofol | Each 2 hours for 48 hours
  In mg
Total dose of fentanyl | Each 2 hours for 48 hours
  In mcg
SAS (Sedation Agitation Scale) | Each 2 hours for 48 hours
  The scale evaluates sedation and agitation of a patient, thus the name is "Sedation Agitation Scale". The total range goes from 1 to 7, where: 1 is Unarousable, 2 is Very Sedated, 3 is Sedated, 4 is Calm and Cooperative, 5 is Agitated, 6 is Very Agitated, and 7 is Dangerous Agitation. If clinical indication is a deep sedation, then the patient must reach a SAS 1-2. If clinical indication is a light sedation, then the patient must reach a SAS 3-4. Scores of 5, 6 and 7 must be avoided with drugs.
SEF95 | Each 2 hours for 48 hours
  Spectral Edge Frequency 95
Mean Arterial Pressure | Each 2 hours for 48 hours
  In mmHg
Plasma triglyceride levels | 24 hours and 48 hours
  Central laboratory
Plasma lactate concentration | 24 hours and 48 hours
  Central laboratory
Duration of mechanical ventilation | Up to 30 days
  Since the beginning of the protocol
Stay in intensive unit care | Up to 30 days
  Since the beginning of the protocol
Wake up after stopping the infusion of propofol | Up to 48 hours
Delirium | Up to 10 days
  Evaluated with CAM-ICU twice a day during the stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Antonello Penna, MD/PhD, Principal Investigator — University of Chile; Rodrigo Gutiérrez, MD, Principal Investigator — University of Chile; Felipe Maldonado, MD, Principal Investigator — University of Chile; José Ignacio Egaña, MD/PhD, Principal Investigator — University of Chile; Eduardo Tobar, MD, Principal Investigator — University of Chile; Verónica Rojas, Nurse/MSc, Principal Investigator — University of Chile
Locations (2):
- Chile (2):
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM